CLINICAL TRIAL: NCT03118856
Title: Real-time Assessment of the Histology of Colorectal Polyps Using Electronic Chromoendoscopy
Brief Title: Electronic Chromoendoscopy for Polyp Characterization
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: TR-001
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HD-WLE: Intervention: Prediction of polyp histology with HD-WLE
  Interventions: Diagnostic Test: Prediction of Histology
- EC: Intervention: Prediction of polyp histology with EC
  Interventions: Diagnostic Test: Prediction of Histology

INTERVENTIONS:
Diagnostic Test: Prediction of Histology — The accuracy of predicting the histology of colorectal polyps will be assessed with HD-WLE and EC

SUMMARY:
To assess the accuracy of predicting histology of colorectal polyps with electronic chromoendoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing screening or surveillance colonoscopy
* written informed consent

Exclusion Criteria:

* inadequate bowel preparation
* polyposis syndromes
* history of colectomy
* use of anticoagulants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing screening or surveillance colonoscopy
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of predicting histology with EC | 1 year
  Polyps will be visualized in white-light and the location and size will be noted. Afterwards, electronic chromoendoscopy will be used to visualize and enhance the mucosal vascular pattern and the mucosal surface pattern morphology of the polyp. The endoscopist will then make a real time assessment of each polyp according to size, shape, Paris classification and surface characteristics including pit pattern and mucosal vascular pattern morphology, colour, and type of depression. Further, a level of confidence (high or low) will be made for the real time histology prediction. Finally, all polyps will be removed using standard techniques and processed for pathological evaluation and real time and histological results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Rath, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Germany